CLINICAL TRIAL: NCT02350777
Title: Phase II Trial of T-cell Depleted Hematopoietic Stem Cell Boosts Without Conditioning for Poor Marrow Graft Function Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: T-cell Depleted Hematopoietic Stem Cell Boosts Without Conditioning for Poor Marrow Graft Function Following Allogeneic Hematopoietic Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-228
Record Dates: First submitted 2015-01-21; First posted 2015-01-30 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2017-10

CONDITIONS: Hematopoietic Stem Cell Transplant; Poor Marrow Graft Function
Keywords: T-cell Depleted Hematopoietic Stem Cell; Allogeneic Hematopoietic Stem Cell Transplantation; CliniMACS Cell Selection System; 14-228; HSCT

ARMS (2):
- active infection and/or organ compromise or GVHD. (Experimental): This protocol includes two single-arm phase II trials to assess the efficacy and confirm the safety of administration of TCD stem cell boost or bone marrow (BM) HPC (M) boost from the original donor for patients with poor graft function after allogeneic hematopoietic stem cell transplantation.
  Interventions: Procedure: Donor peripheral blood progenitor cells: stimulation, harvesting, isolation and T-cell depletion; Device: CliniMACS Cell Selection System
- active infection, active or controlled GVHD &/or organ compro (Experimental): This protocol includes two single-arm phase II trials to assess the efficacy and confirm the safety of administration of TCD stem cell boost or bone marrow (BM) HPC (M) boost from the original donor for patients with poor graft function after allogeneic hematopoietic stem cell transplantation.
  Interventions: Procedure: Donor peripheral blood progenitor cells: stimulation, harvesting, isolation and T-cell depletion; Device: CliniMACS Cell Selection System

INTERVENTIONS:
Procedure: Donor peripheral blood progenitor cells: stimulation, harvesting, isolation and T-cell depletion — For related donors, beginning 5-6 days before the day of HPC(A) or HPC (M) TCD boost infusion, the normal donor will receive GCSF per institutional guidelines. On the fifth and sixth days of this course of G-CSF, the donor will undergo daily leukapheresis designed to provide a minimum of 5x10^6 CD34+ cells/kg of the transplant recipient's weight. For unrelated donors, the G-CSF will be administered and the leukapheresis obtained according to the National Marrow Donor Program protocol IND, and institutional guidelines. Mononuclear cell fractions (i.e., CD34+ cells) collected on the fourth and fifth days will be pooled.
Device: CliniMACS Cell Selection System

SUMMARY:
The purpose of this study is to see if giving the patient stem cells their original donor (boost) after removing the T cells (T cell depleted- TCD boost) without further chemotherapy. The investigators want to see if this can improve bone marrow function. This would also improve the patients white blood counts, red blood counts and platelets. This may make the patients chances of improving and surviving better. The investigators will also be looking at the short term side effects and risks of the TCD boost.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with PGF are candidates for this trial.
* Patients who underwent transplant at another facility and suffer from PGF will be eligible as well as long as a donor is available. PGF can be primary (no counts recovery after the preparative regimen) or secondary (cytopenia after engraftment has occurred).
* Patients with auto-immune cytopenia with auto antibodies to neutrophils or platelets or positive Coombs test that did not respond to immunosuppressive agents within 3 months from initiation of therapy are eligible as well.
* Persistent cytopenia requiring growth factors and/or blood products AND evidence of hypocellular BM (<25%). Persistent cytopenia (at least 4 weeks period) is defined by presence of TWO of the following:

  1. ANC <1.0x10^9/L without filgrastim support or any ANC value that requires recurrent support by filgrastim (administered at least once a week).
  2. Plt<50x10^9/L
  3. Hb<8 or PRBC transfusion dependent (once every 2 weeks or more) with reticulocyte count of < 40x10^9/L.

This criteria for persistent cytopenia and hypocellular bone marrow does not apply to patients with auto-immune cytopenia, ONLY PGF patients

* Full donor myeloid chimerism. Patients after T cell depletion transplant can have a significant mixed T cell chimerism and this can affect the testing of marrow chimerism. In this case, the neutrophil chimerism will be used to determine eligibility for this trial. Patients will be excluded if neutrophils are less than 90% donor cells; a higher percentage of host cells could be due to relapse or impending relapse.
* Age: pediatrics and adults patients. No age exclusion.
* Each patient must be willing to participate as a research subject and must sign an informed consent form.
* For infections and end organs related criteria (at time of TCD boost administration) see table in protocol.

Exclusion Criteria:

Patients will be excluded from the trial if at time of enrollment:

* Evidence of relapsed disease by morphologic, cytogenetic or molecular diagnostic tools.
* Hypersplenism documented by imaging study (US or CT)
* Pregnant women
* Patient who underwent TCD boost without counts recovery and are considered for another TCD boost will be treated off protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roni Tamari, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- No Active Infection and/or Organ Compromise or GVHD.; Active Infection, Active or Controlled GVHD &/or Organ Compro: This protocol includes two single-arm phase II trials to assess the efficacy and confirm the safety of administration of TCD stem cell boost or bone marrow (BM) HPC (M) boost from the original donor for patients with poor graft function after allogeneic hematopoietic stem cell transplantation.
Period: Overall Study
Arm/Group | No Active Infection and/or Organ Compromise or GVHD. | Active Infection, Active or Controlled GVHD &/or Organ Compro
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Active Infection and/or Organ Compromise or GVHD. | Active Infection, Active or Controlled GVHD &/or Organ Compro | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 54 [50 to 58] | 50 [45 to 55] | 52 [45 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Blood Counts Recovery (Response Will be Defined by Stable Blood Counts (ANC>1000, Hb>8 With Absolute Reticulocyte Count>20x10^9/L ,and Plt>50,000) Without Support of Blood Product Transfusions and/or Growth Factors.
Description: will be documented by CBC checks every 2 weeks. Response will be defined by stable blood counts (ANC>1000, Hb>8 with absolute reticulocyte count>20x10^9/L ,and Plt>50,000) without support of blood product transfusions and/or growth factors.
Time Frame: 1 year
Population: No data were collected
Arm/Group | No Active Infection and/or Organ Compromise or GVHD. | Active Infection, Active or Controlled GVHD &/or Organ Compro
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | No Active Infection and/or Organ Compromise or GVHD. | Active Infection, Active or Controlled GVHD &/or Organ Compro
All-Cause Mortality (participants affected / at risk) | 1/2 | 1/2
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No Active Infection and/or Organ Compromise or GVHD. (N=2) | Active Infection, Active or Controlled GVHD &/or Organ Compro (N=2)
Pericardial tamponade (Cardiac disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Active Infection and/or Organ Compromise or GVHD. (N=2) | Active Infection, Active or Controlled GVHD &/or Organ Compro (N=2)
Creatinine increased (Investigations) | 2 (6) | 0
Pericardial tamponade (Cardiac disorders) | 1 | 0
Alkaline phosphatase increased (Investigations) | 0 | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (3) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT02350777/Prot_SAP_000.pdf